CLINICAL TRIAL: NCT04802759
Title: A Phase Ib/II, Open-Label, Multicenter, Randomized Umbrella Study Evaluating the Efficacy and Safety of Multiple Treatment Combinations in Patients With Breast Cancer (MORPHEUS-BREAST CANCER)
Brief Title: A Study Evaluating the Efficacy and Safety of Multiple Treatment Combinations in Participants With Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO42867; 2020-004889-19 (EudraCT Number); 2023-507495-48-00 (EU CTIS Number)
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Inoperable, Locally Advanced or Metastatic, ER-positive Breast Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — giredestrant; abemaciclib; ipatasertib; inavolisib; ribociclib; Everolimus; pertuzumab; Trastuzumab; palbociclib; atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (16):
- Cohort 1: Giredestrant Monotherapy (Active Comparator)
  Interventions: Drug: Giredestrant
- Cohort 1: Giredestrant + Abemaciclib (Experimental)
  Interventions: Drug: Giredestrant; Drug: Abemaciclib
- Cohort 1: Giredestrant + Ipatasertib (Experimental)
  Interventions: Drug: Giredestrant; Drug: Ipatasertib
- Cohort 1: Giredestrant + Inavolisib (Experimental)
  Interventions: Drug: Giredestrant; Drug: Inavolisib
- Cohort 1: Giredestrant + Ribociclib (Experimental)
  Interventions: Drug: Giredestrant; Drug: Ribociclib
- Cohort 1: Giredestrant + Everolimus (Experimental)
  Interventions: Drug: Giredestrant; Drug: Everolimus
- Cohort 1: Giredestrant + Samuraciclib (Experimental)
  Interventions: Drug: Giredestrant; Drug: Samuraciclib
- Cohort 1: Giredestrant + Atezolizumab (Experimental)
  Interventions: Drug: Giredestrant; Drug: Atezolizumab
- Cohort 1: Giredestrant + Abemaciclib + Atezolizumab (Experimental)
  Interventions: Drug: Giredestrant; Drug: Abemaciclib; Drug: Atezolizumab
- Cohort 1: Giredestrant + Inavolisib (ESR1m enriched) (Experimental): ESR1m stands for estrogen receptor mutation.
  Interventions: Drug: Giredestrant; Drug: Inavolisib
- Cohort 2: Giredestrant + PH FDC SC (Active Comparator)
  Interventions: Drug: Giredestrant; Drug: PH FDC SC
- Cohort 2: Giredestrant + PH FDC SC + Abemaciclib (Experimental)
  Interventions: Drug: Giredestrant; Drug: Abemaciclib; Drug: PH FDC SC
- Cohort 2: Giredestrant + PH FDC SC + Palbociclib (Experimental)
  Interventions: Drug: Giredestrant; Drug: PH FDC SC; Drug: Palbociclib
- Cohort 3: Giredestrant + Inavolisib + Palbociclib (Experimental)
  Interventions: Drug: Giredestrant; Drug: Inavolisib; Drug: Palbociclib
- Cohort 3: Giredestrant + Inavolisib + Abemaciclib (Experimental)
  Interventions: Drug: Giredestrant; Drug: Abemaciclib; Drug: Inavolisib
- Cohort 3: Giredestrant + Inavolisib + Ribociclib (Experimental)
  Interventions: Drug: Giredestrant; Drug: Inavolisib; Drug: Ribociclib

INTERVENTIONS:
Drug: Giredestrant — 30 milligrams (mg) orally once a day (during each 28-day cycle or 21-day cycle, depending on the regimen) until unacceptable toxicity or disease progression
  Other Names: GDC-9545; RO7197597; RG6171
Drug: Abemaciclib — 150 mg orally twice a day (during each 28-day cycle or 21-day cycle, depending on the regimen) until unacceptable toxicity or disease progression
  Other Names: Verzenio™
  Arms: Cohort 1: Giredestrant + Abemaciclib; Cohort 1: Giredestrant + Abemaciclib + Atezolizumab; Cohort 2: Giredestrant + PH FDC SC + Abemaciclib; Cohort 3: Giredestrant + Inavolisib + Abemaciclib
Drug: Ipatasertib — 400 mg orally once a day on Days 1-21 of each 28-day cycle until unacceptable toxicity or disease progression
  Other Names: GDC-0068; RO5532961; RG7440
  Arms: Cohort 1: Giredestrant + Ipatasertib
Drug: Inavolisib — 9 mg orally once a day during each 28-day cycle until unacceptable toxicity or disease progression
  Other Names: ITOVEBI™; GDC-0077; RO7113755; RG6114
  Arms: Cohort 1: Giredestrant + Inavolisib; Cohort 1: Giredestrant + Inavolisib (ESR1m enriched); Cohort 3: Giredestrant + Inavolisib + Abemaciclib; Cohort 3: Giredestrant + Inavolisib + Palbociclib; Cohort 3: Giredestrant + Inavolisib + Ribociclib
Drug: Ribociclib — 600 mg orally once a day on Days 1-21 of each 28-day cycle until unacceptable toxicity or disease progression
  Other Names: Kisqali®
  Arms: Cohort 1: Giredestrant + Ribociclib; Cohort 3: Giredestrant + Inavolisib + Ribociclib
Drug: Everolimus — 10 mg orally once a day during each 28-day cycle until unacceptable toxicity or disease progression
  Other Names: Afinitor®
  Arms: Cohort 1: Giredestrant + Everolimus
Drug: Samuraciclib — 360 mg orally once a day during each 28-day cycle until unacceptable toxicity or disease progression
  Other Names: ICEC0942; CT7001
  Arms: Cohort 1: Giredestrant + Samuraciclib
Drug: PH FDC SC — On Day 1 of Cycle 1 (1 cycle is 21 days), pertuzumab and trastuzumab fixed-dose combination for subcutaneous use (PH FDC SC) will be administered SC as a fixed dose formulation of 1200 mg pertuzumab, 600 mg trastuzumab, and 30,000 units hyaluronidase. On Day 1 of Cycles 2 and beyond, PH FDC SC will be administered SC once every 21 days as a fixed dose of 600 mg pertuzumab, 600 mg trastuzumab, and 20,000 units hyaluronidase.
  Other Names: Pertuzumab, Trastuzumab, and Hyaluronidase-zzxf; PHESGO™; RO7198574; RG6264
  Arms: Cohort 2: Giredestrant + PH FDC SC; Cohort 2: Giredestrant + PH FDC SC + Abemaciclib; Cohort 2: Giredestrant + PH FDC SC + Palbociclib
Drug: Palbociclib — 125 mg orally once a day on Days 1-21 during each 28-day cycle until unacceptable toxicity or disease progression
  Other Names: Ibrance®
  Arms: Cohort 2: Giredestrant + PH FDC SC + Palbociclib; Cohort 3: Giredestrant + Inavolisib + Palbociclib
Drug: Atezolizumab — 840 mg by intravenous (IV) infusion on Days 1 and 15 each 28-day cycle.
  Other Names: Tecentriq®; RO5541267; RG7446
  Arms: Cohort 1: Giredestrant + Abemaciclib + Atezolizumab; Cohort 1: Giredestrant + Atezolizumab

SUMMARY:
This is a Phase Ib/II, open-label, multicenter, randomized umbrella study in participants with breast cancer. The study is designed with the flexibility to open new treatment arms as new treatments become available, close existing treatment arms that demonstrate minimal clinical activity or unacceptable toxicity, or modify the patient population.

Cohort 1 will focus on participants with inoperable, locally advanced or metastatic, estrogen receptor-positive (ER+), HER2-negative breast cancer who had disease progression during or following treatment with a cyclin-dependent kinase 4/6 inhibitor (CDK4/6i; e.g., palbociclib, ribociclib, abemaciclib) in the first- or second-line setting.

Cohort 2 will focus on inoperable, locally advanced or metastatic, ER+, HER2-positive breast cancer with previous progression to standard-of-care anti-HER2 therapies, of which one was a trastuzumab-and-taxane-based systemic therapy (including in the early setting if recurrence occurred within 6 months of finishing adjuvant therapy) and one was a HER2-targeting antibody-drug conjugate (ADC; e.g., ado-trastuzumab emtansine or trastuzumab-deruxtecan) or a HER2-targeting tyrosine kinase inhibitor (TKI; e.g., tucatinib, lapatinib, pyrotinib, or neratinib).

Cohort 3 will focus on inoperable, locally advanced or metastatic, ER+, HER2-negative, PIK3CA-mutated breast cancer with resistance to adjuvant endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Cohort 1 (Stage 1 [and Stage 2, only where indicated]):

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Documented estrogen receptor-positive (ER+) tumor
* Patients for whom endocrine therapy is recommended and treatment with cytotoxic chemotherapy is not indicated at time of entry into the study, as per national or local treatment guidelines
* Radiologic/objective evidence of recurrence or progression after the most recent systemic therapy for breast cancer
* Disease progression during or after first- or second-line hormonal therapy for locally advanced or metastatic disease (note: at least one line of therapy must have contained a CDK4/6i administered for a minimum of 8 weeks prior to disease progression.)
* Postmenopausal status for women
* Life expectancy ≥3 months
* Availability of a representative tumor specimen that is suitable for biomarker evaluation via central testing
* Prior fulvestrant therapy is allowed
* Stages 1 and 2: Measurable disease (at least one target lesion) according to RECIST v1.1
* Stages 1 and 2: Adequate hematologic and end-organ function
* Stages 1 and 2: Stable anticoagulant regimen for patients receiving therapeutic anticoagulation

Inclusion Criteria for Cohort 2 (Stage 1 [and Stage 2, only where indicated]):

* ECOG Performance Status of 0 or 1
* Histologically or cytologically confirmed and documented adenocarcinoma of the breast with metastatic or locally advanced disease not amenable to curative resection
* ER+, HER2-positive breast cancer
* Postmenopausal status for women
* Life expectancy ≥3 months
* Willingness to have a representative tumor specimen that is suitable for biomarker evaluation via central testing submitted, if available
* Prior endocrine therapy in the advanced setting allowed, including fulvestrant if given more than 28 days prior to randomization, but excluding other selective estrogen receptor degraders (SERDs)
* Stages 1 and 2: Measurable disease (at least one target lesion) according to RECIST v1.1
* Stages 1 and 2: Baseline left ventricular ejection fraction (LVEF) ≥50% as measured by ECHO or MUGA scans
* Stages 1 and 2: Adequate hematologic and end-organ function
* Stages 1 and 2: Stable anticoagulant regimen for patients receiving therapeutic anticoagulation

Inclusion Criteria for Cohorts 1 and 2 (Stage 2):

* Ability to initiate Stage 2 treatment within 3 months after experiencing unacceptable toxicity, disease progression as determined by the investigator according to RECIST v1.1, or loss of clinical benefit as determined by the investigator, provided that a Stage 2 slot is available and patient meets eligibility criteria for Stage 2
* Availability of a tumor specimen from a biopsy performed upon discontinuation of Stage 1 because of unacceptable toxicity to drugs, disease progression as determined by the investigator according to RECIST v1.1, or loss of clinical benefit as determined by the investigator

Inclusion Criteria for Cohort 3:

* Measurable disease (at least one target lesion) according to RECIST v1.1
* ECOG Performance Status of 0 or 1
* Documented ER+ tumor
* Patients for whom endocrine therapy is recommended and treatment with cytotoxic chemotherapy is not indicated at time of entry into the study, as per national or local treatment guidelines
* Histologically or cytologically confirmed and documented adenocarcinoma of the breast that is locally advanced or metastatic and is not amenable to surgical or radiation therapy with curative intent
* Patients must have progressed during adjuvant endocrine treatment or within 12 months of completing adjuvant endocrine therapy with an aromatase inhibitor or tamoxifen. If a CDK4/6i was included as part of neoadjuvant or adjuvant therapy, progression event must be >12 months since completion of CDK4/6i portion of neoadjuvant or adjuvant therapy.
* Postmenopausal status for women (including women on or starting luteinizing hormone-releasing hormone [LHRH] agonist for ovarian suppression prior to randomization)
* Life expectancy ≥6 months
* Adequate hematologic and end-organ function
* Evidence of an eligible PIK3CA mutation based on pre-existing test results (i.e., previously obtained as part of clinical practice) from blood or tumor tissue. If pre-existing test results are not available, submission of a freshly collected pretreatment blood sample to determine PIK3CA mutation status at a central testing site with the FoundationOne Liquid® CDx assay is required.

Exclusion Criteria:

General Exclusion Criteria for all Treatment Arms in Stage 1, Cohorts 1 and 2 (unless only applicable to one cohort, as indicated):

* Prior treatment with any of the protocol-specified study treatments
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Systemic treatment for breast cancer within 2 weeks of Cycle 1, Day 1 or 5 half-lives of the drug prior to Cycle 1, Day 1
* Treatment with strong CYP3A4 inhibitors or inducers within 14 days or 5 drug elimination half-lives (whichever is longer) prior to randomization
* Adverse events from prior anti-cancer therapy that have not resolved to Grade ≤1 or better, with the exception of alopecia of any grade and Grade ≤2 peripheral neuropathy
* Eligible only for the control arm
* Prior allogeneic stem cell or solid organ transplantation
* Major surgical procedure other than for diagnosis within 4 weeks prior to initiation of study treatment or anticipation of need for a major surgical procedure during the course of the study
* History of malignancy other than breast cancer within 2 years prior to screening, with the exception of those with a negligible risk of metastasis or death
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Uncontrolled tumor-related pain
* Uncontrolled or symptomatic hypercalcemia
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* History of leptomeningeal disease
* Active tuberculosis
* Severe infection within 4 weeks prior to initiation of study treatment
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography scan
* Active cardiac disease or history of cardiac dysfunction
* Positive HIV test at screening or at any time prior to screening
* Active Hepatitis B or Hepatitis C virus infection
* Active inflammatory bowel disease, chronic diarrhea, short bowel syndrome, or major upper gastrointestinal (GI) surgery, including gastric resection, potentially affecting enteral absorption
* Known allergy or hypersensitivity to any of the study drugs or any of their excipients
* Cohort 1 only: Known HER2-positive breast cancer
* Cohort 1 only: Concurrent hormone replacement therapy
* Cohort 1 only: Prior treatment with cytotoxic chemotherapy for metastatic breast cancer (with the exception of single agent capecitabine, which will count as a single line of therapy)
* Cohort 2 only: Dyspnea at rest due to complications of advanced malignancy, or other disease requiring continuous oxygen therapy
* Cohort 2 only: Current chronic daily treatment (continuous for >3 months) with corticosteroids (dose of 10 mg/day methylprednisolone equivalent), excluding inhaled steroids

Additional Exclusion Criteria for Giredestrant + Abemaciclib Arm and Giredestrant + Abemaciclib + Atezolizumab Arm (Cohort 1, Stage 1):

* Interstitial lung disease or severe dyspnea at rest or requiring oxygen therapy
* History of major surgical resection involving the stomach or small bowel, or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea
* History of syncope of cardiovascular etiology, ventricular arrhythmia, or sudden cardiac arrest

Additional Exclusion Criteria for Giredestrant + Ipatasertib Arm (Cohort 1, Stage 1):

* Prior treatment with an Akt inhibitor
* Inability to swallow medication or malabsorption condition that would alter the absorption of orally administered medications
* Grade ≥2 uncontrolled or untreated hypercholesterolemia or hypertriglyceremia
* History of Type 1 or Type 2 diabetes mellitus requiring insulin
* History or presence of an abnormal electrocardiogram (ECG) that is clinically significant in the investigator's opinion

Additional Exclusion Criteria for the Giredestrant + Inavolisib and Giredestrant + Inavolisib (ESR1m enriched) Arms (Cohort 1, Stage 1):

* Prior treatment with any PI3K, Akt, or mTOR inhibitor, or any agent whose mechanism of action is to inhibit the PI3K/Akt/mTOR pathway
* Type 2 diabetes requiring ongoing systemic treatment at the time of study entry; or any history of Type 1 diabetes
* Fasting glucose ≥126 mg/dL or ≥7.0 mmol/L and HbA1c ≥5.7% (or HbA1c ≥6.4% for the ESR1m enriched Arm only)
* Any concurrent ocular or intraocular condition, excluding baseline cataracts, that, in the opinion of the investigator, would require medical or surgical intervention during the study period to prevent or treat vision loss
* Active inflammatory or infectious conditions in either eye or history of idiopathic or autoimmune-associated uveitis in either eye
* Symptomatic active lung disease, including pneumonitis
* Inability to confirm biomarker eligibility based on valid results from either central testing of blood or local testing of blood or tumor tissue that documents one of the protocol-defined PIK3CA mutations
* ESR1m enriched Arm only: Inability to determine ESR1 mutation status based on valid results from either central testing of blood or from pre-existing test results (from blood or tumor tissue) that confirm the presence of an ESR1 mutation. While patients who have tumors without detectable ESR1 mutation may be enrolled in this arm, a pre-existing test with no detectable ESR1m result is not acceptable for enrollment, and the participant in this case must submit a sample for central testing.

Additional Exclusion Criteria for Giredestrant + Ribociclib Arm (Cohort 1, Stage 1):

* Currently receiving or has received systemic corticosteroids ≤2 weeks prior to starting trial treatment
* Impairment of GI function or GI disease that may significantly alter the absorption of the oral trial treatments

Additional Exclusion Criteria for Giredestrant + Samuraciclib Arm (Cohort 1, Stage 1):

* Prior treatment with mTOR inhibitor
* Receipt of systemic corticosteroids (at a dose >10 mg prednisone/day or equivalent) within 14 days before the first dose of samuraciclib
* Active bleeding diatheses
* History of hemolytic anemia or marrow aplasia
* Receipt of a live-virus vaccination within 28 days or less of planned treatment start

Additional Exclusion Criteria for Giredestrant + Atezolizumab-Containing Arms (Cohort 1, Stage 1):

* Active or history of autoimmune disease or immune deficiency
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab
* Treatment with systemic immunostimulatory agents within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or recombinant human antibodies
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Pregnant or breastfeeding, or intending to become pregnant during study treatment or within 5 months for atezolizumab

Additional Exclusion Criteria for Giredestrant + PH FDC SC + Abemaciclib Arm (Cohort 2, Stage 1):

* Interstitial lung disease or severe dyspnea
* History of major surgical resection involving the stomach or small bowel, preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea, or a condition that may significantly alter the absorption of the oral trial treatments
* History of syncope of cardiovascular etiology, ventricular arrhythmia, or sudden cardiac arrest

Additional Exclusion Criteria for Giredestrant + PH FDC SC + Palbociclib Arm (Cohort 2, Stage 1):

* History of major surgical resection involving the stomach or small bowel, preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea, or a condition that may significantly alter the absorption of the oral trial treatments
* Interstitial lung disease or severe dyspnea

Exclusion Criteria for Cohort 3:

* Known HER2-positive breast cancer
* Prior treatment with any SERD (e.g., fulvestrant, novel oral), proteolysis targeting chimera, complete ER antagonist (CERAN), or novel SERM (other than tamoxifen, toremifene)
* Prior treatment with any PI3Kalpha (PIK3CA gene product), AKT or mTOR inhibitor
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Treatment with strong CYP3A4 inhibitors or inducers within 14 days or 5 drug elimination half-lives (whichever is longer) prior to randomization
* Adverse events from prior anti-cancer therapy that have not resolved to Grade ≤1 or better, with the exception of alopecia of any grade and Grade ≤2 peripheral neuropathy
* Major surgical procedure within 4 weeks prior to initiation of study treatment or anticipation of need for a major surgical procedure during the course of the study
* History of malignancy other than breast cancer within 2 years prior to screening, with the exception of those with a negligible risk of metastasis or death
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Uncontrolled tumor-related pain
* Uncontrolled or symptomatic hypercalcemia
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* History of leptomeningeal disease
* Severe infection within 4 weeks prior to initiation of study treatment
* Treatment for clinically significant infection with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography scan
* Active cardiac disease or history of cardiac dysfunction
* Positive HIV test at screening or at any time prior to screening
* Active Hepatitis B or Hepatitis C virus infection
* Active inflammatory bowel disease, chronic diarrhea, short bowel syndrome, or major upper gastrointestinal (GI) surgery, including gastric resection, potentially affecting enteral absorption
* Known allergy or hypersensitivity to any of the study drugs or any of their excipients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2029-05-30 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Objective Response, Defined as a Complete or Partial Response, as Determined by the Investigator According to Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1) | From Baseline until disease progression (up to 6 years)
Number of Participants with Adverse Events, Severity Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE v5.0) | From Baseline until 30 days after the last dose of study drug (up to 6 years)

SECONDARY OUTCOMES:
Progression-Free Survival, as Determined by the Investigator According to RECIST v1.1 | From randomization to the date of the first recorded occurrence of disease progression or death from any cause, whichever occurs first (up to 6 years)
Disease Control Rate, Defined as the Percentage of Participants with Stable Disease for ≥12 Weeks or a Complete or Partial Response, as Determined by the Investigator According to RECIST v1.1 | From Baseline until disease progression (up to 6 years)
Clinical Benefit Rate, Defined as the Percentage of Participants with Stable Disease for ≥24 Weeks or with Confirmed Complete or Partial Response, as Determined by the Investigator According to RECIST v1.1 | From Baseline until disease progression (up to 6 years)
Overall Survival | From randomization to death from any cause (up to 6 years)
Duration of Response, as Determined by the Investigator According to RECIST v1.1 | From first occurrence of a document objective response to the first date of recorded disease progression or death from any cause, whichever occurs first (up to 6 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (31):
- United States (11):
  - City of Hope, Duarte, California
  - University of California, San Francisco (UCSF), San Francisco, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Santa Monica, California
  - Stanford Cancer Institute (SCI), Stanford, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Regional Cancer Care Associates LLC (RCCA) - Freehold Location, Freehold, New Jersey
  - Regional Cancer Care Associates LLC ? Howell Division, Howell Township, New Jersey
  - Levine Cancer Institute, Charlotte, North Carolina
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - West Cancer Center, Germantown, Tennessee
- Australia (4):
  - Flinders Medical Centre, Bedford Park, South Australia
  - Peninsula Health-Frankston Hospital, Frankston, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Linear Clinical Research Limited, Nedlands, Western Australia
- Israel (7):
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Rambam Medical Center, Haifa
  - Hadassah Ein Karem Hospital, Jerusalem
  - Rabin MC, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assuta Medical Centers, Tel Aviv
- South Korea (5):
  - National Cancer Center, Goyang-si
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (4):
  - Hospital Universitario Vall d Hebron, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Centro Integral Oncológico Clara Campal Ensayos Clínicos START, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing